CLINICAL TRIAL: NCT03882567
Title: Effectiveness of Electro Neuro Adaptive Regulator on Pain, Disability and Central Sensitization in Patients With Fibromyalgia
Brief Title: Effectiveness of Electro Neuro Adaptive Regulator in Patients With Fibromyalgia
Acronym: SCENAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, Professor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 03/2015
Record Dates: First submitted 2018-09-04; First posted 2019-03-20 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Fibromyalgia
Keywords: visual analogue scale; conditioned pain modulation; disability; pressure pain threshold; temporal summation
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electro Neuro adaptative Regulator (Experimental): 8 SCENAR sessions (twice a week) (30 min of duration) following the protocols for treatment several points in the body
  Interventions: Other: Electro Neuro adaptative Regulator
- Sham Electro Neuro adaptative Regulator (Sham Comparator): 8 Sham SCENAR sessions (twice a week) (30 min of duration), following the same protocol tan experimental group but the machine will be turn off 30 seconds after starting on the treatment.
  Interventions: Other: Electro Neuro adaptative Regulator

INTERVENTIONS:
Other: Electro Neuro adaptative Regulator — The SCENAR device has been previously described and generates high-amplitude, pulsed, damped biphasic sinusoidal current that is delivered to the tissue via a pair of concentric electrodes placed in direct contact with the target area. The intensity of the interactive waveform adjusts in response to changes in skin impedance
  Other Names: InterX

SUMMARY:
Background: There is evidence linking conditioned pain modulation (CPM) deficiency with musculoskeletal pain syndromes such as fibromyalgia, Evidence shows that different physical therapies could activation situations of chronic pain there is no activation of CPM.

Objectives: The purpose of this study is to measure the CPM response and determine whether Electro Neuro Adaptative Regulator in patients with Fibromyalgia is effective in the improvement of CPM, TS, pain intensity, disability.

Design: Double-blind, randomized placebo clinical trial. Methods: Patients with fibromyalgia will be randomly allocated into two groups: the Electro Neuro Adaptative Regulator group (SCENAR) or the sham technique (ST) group.

Main outcomes measures: Pain intensity (with visual analogue scale, Conditioned Pain Modulation (CPM), Temporal Summation (TS) and Pressure Pain Thresholds (PPT´s) were the primary outcomes and will be assessed at baseline and at 3-months follow-up. Secondary outcome measures were the Fibromyalgia Impact Questionnaire to measure disability, Pain Catastrophizing Scale and the Pain Anxiety Symptoms Scale, Beck Depression Inventory, Jenkins Sleep Scale. Questionnaire of quality of life SF36.

Participants will be selected if they met the following inclusion criteria: (a) fulfilled the 1990 and 2010 American College of Rheumatology classification criteria for FM; (b) reported an average pain intensity ≥ 4 on a 0 to 10 cm visual analogue scale during the previous week to study commencement; (c) were on stable doses of medication for FM ≥ 4 weeks; and (d) were aged between 18 and 65 years.

ELIGIBILITY:
Inclusion Criteria:

1. . American College of Rheumatology classification criteria for Fibromyalgia.
2. . reported average pain intensity ≥ 4 on a 0 to 10 cm visual analogue scale based on 1 week of daily pain diaries;
3. on stable doses of medications for FM ≥ 4 weeks.

Exclusion Criteria:

* Patients will be excluded from enrolment if: (1) they suffer from an inflammatory rheumatic conditions; (2) have a planned elective surgery during the study period; (3) have ongoing unresolved disability claims; (4) experience symptoms of bipolar disorder, major depressive disorder, panic disorder, or psychosis; (5) do not speak Spanish fluently.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Numerical pain ranting Scale | Change from Baseline of pain intensity at 3 months
  The patients will be asked to assess the subjective pain intensity of the painful in whole body by to marking the level of pain on the scale. Pain intensity was measured with the NRS of 11 points (interval from 0 to 10), where 0 corresponds to no pain, and 10 corresponds to the worst pain imaginable.
Fibromyalgia Impact Questionnaire (FIQ) | Change from Baseline of Fibromyalgia impact questionnaire at 3 months
  The FIQ, which is a validated self-reported questionnaire to measure multidimensional function/health-related quality of life, will be used.Scores in the FIQ range from 0 to 100, An improvement greater than 30% in the FIQ total score has been identified in clinical trials as sensitive to identify a positive response to treatment.

SECONDARY OUTCOMES:
Conditioned pain modulation | Change from Baseline of CPM at 3 months
  After an interval of 5 minutes CPM was assessed by replicating the TS assessment associated with a conditioning stimulus for eliciting CPM. The conditioning stimulus was an occlusion cuff at the left arm inflated, at a rate of 20 mmHg/s until the subject reports "the first sensation of pain". Acquired pressure at this point remained for 30 seconds. The subject described the intensity of pain, because of occlusion in the arm, on a verbal numerical rating scale (0 = no pain and 10 = worst possible pain). Then cuff inflation was increased or decreased until the intensity of pain will be 3/10 in verbal rating scale
Mechanical Hyperalgesia | Change from Baseline of PPT at 3 months
  Pressure Pain Thresholds (PPTs) were assessed using algometry in the thumb (dorsal aspect of the distal phalanx). The PPT is defined as the lowest pressure that, using standardized testing conditions, needs to be applied to cause the slightest sensation of pain. It is a reliable and widely used measure
Temporal Summation | Change from Baseline of TS at 3 months
  The degree of TS or wind-up will be evaluated in response to 10 applications (pulses) of the algometer, with an approximate rate of pressure increase of 2 Kg/s, at the previously defined PPT at the dorsal surface of the right-hand middle finger midway between the first and second distal joints, and at the middle of the right-hand side upper trapezius belly. Participants were asked to rate the intensity and unpleasantness of the pain intuitively of the first, fifth, and tenth pulse on a numeric pain rating scale.
Pain Catastrophizing | Change from Baseline of pain catastrophizing at 3 months
  The Spanish version of the Pain Catastrophizing Scale (PCS) was used to assess catastrophic thoughts about pain, which has shown appropriate psychometric properties.
State Trait Anxiety Inventory | Change from Baseline of Anxiety at 3 months
  All participants will complete the Spanish version of the trait subscale of the State Trait Anxiety Inventory (STAI-T). The STAI-T has been found to possess adequate reliability (alpha coefficients of 0.93, test-retest reliability of 0.80) and validity.
Beck Depression Inventory (BDI) | Change from Baseline of Depression symptoms at 3 months
  The level of depressive symptomatology was measured by the Spanish version of the Beck Depression Inventory (BDI-II); a self-report measure that assesses affective, cognitive and somatic symptoms of depression.
Tampa Scale for Kinesiophobia | Change from Baseline of kinesiophobia at 3 months
  Developed by Miller, will be used to assess fear of movement and injury. We'll use the original 17-item version, which has shown good psychometric guarantees
Jenkins Sleep Scale | Change from Baseline of sleep scale at 3 months
  The Jenkins Sleep Scale (JSS) is a 4-item self-report questionnaire designed to measure how often a subject has experienced sleep problems in the past month and has been studied in FM patients and found to be valid, reliable, and able to detect change after treatment.
SF-36. Short Form-36 Health Survey | Change from Baseline of quality of life at 3 months
  The Health related of quality of life will be selected primary outcome. It is a multipurpose, form health survey that includes 36 items taken directly from eight scale scores (physical functioning [PF], role-physical [RP], bodily pain [BP], general health [GH], vitality [VT], social functioning [SF], role-emotional [RE], and mental health [MH]).

CONTACTS AND LOCATIONS:
Overall Officials: Josue Fernández-Carnero, PhD, Study Director — Universidad Rey Juan Carlos
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain